CLINICAL TRIAL: NCT07050758
Title: Pain Reprocessing Therapy for Chronic Widespread Pain - A Randomized Multiple-baseline SCED Trial
Brief Title: Pain Reprocessing Therapy for Chronic Widespread Pain: a SCED Study
Acronym: FOKUS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Kristiania University College (Other)
Responsible Party: Principal Investigator, Dan-Mikael Ellingsen, Professor of Psychology, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025032; 2025032 (Other Grant/Funding Number: Helse Sør-øst)
Record Dates: First submitted 2025-06-12; First posted 2025-07-03 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Pain; Chronic Widespread Pain; Chronic Pain; Fibromyalgia
Keywords: Pain; Chronic widespread pain; Fibromyalgia; Pain reprocessing therapy; SCED; Single-case experimental design
MeSH Terms: conditions — Pain; Chronic Pain; Fibromyalgia

STUDY DESIGN:
Intervention Model Description: The investigators will use a randomized multiple baselines Single-case experimental design. This is a within-subjects design commonly used in SCED studies, in which each participant has a baseline period with a randomized duration (i.e. different participants are assessed for a different number of days prior to treatment onset).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Reprocessing Therapy (Experimental): After a baseline period of 6-14 days (pseudorandomized duration), patients will undergo 9 interventional sessions over a span of 4-6 weeks. This includes an initial consultation with a medical doctor in order to confirm that clinical inclusion criteria are met and exclude potential structural (nociceptive or neuropathic) causes of pain. After this consultation, participants undergo 8 PRT sessions with a clinical psychologist trained in PRT.
  Interventions: Behavioral: Pain Reprocessing Therapy

INTERVENTIONS:
Behavioral: Pain Reprocessing Therapy — Each PRT session will take 45-60 minutes and includes psychoeducation about the association between pain and the brain, mindfulness, and exposure- and acceptance-based concepts. Through PRT, participants will learn about how pain can emerge from 'stuck patterns' in neural circuits in the brain. Through reflections of their own pain experiences, the patient explores evidence for whether this applies to their own pain. Patients will acquire corrective experiences in which their brain "learns" not to respond with pain ("false alarm") in situations that are safe. One central reprocessing exercise is 'somatic tracking', in which participants explore their pain sensations in a context of safety. This includes interoceptive exposures and situational exposures to activities they fear will trigger pain. Exploring these sensations and situations through a lens of safety and curiosity allows the participants to reinterpret bodily sensations previously associated with threat or pain, as safe.

SUMMARY:
Chronic Widespread Pain (CWP) is classified as a Chronic Primary Pain syndrome in the ICD-11 and is considered a major type of nociplastic pain with an estimated prevalence of up to 8-10% in the general population. Many CWP patients experience inadequate treatment and poor symptom management, leaving them prone to disability. Pain Reprocessing Therapy (PRT) is a novel therapy specifically designed to target nociplastic pain with a combination of cognitive, exposure-based, and interoceptively-focused psychotherapy techniques. A recent clinical trial indicated large effects of PRT for chronic back pain, but no studies have yet investigated PRT for CWP. Furthermore, there is little knowledge about how pain and other outcomes change during PRT intervention (between baseline and post-intervention timepoints).

The investigators will use a Single-Case Experimental Design (SCED) to investigate PRT for CWP. Primary outcomes include pain collected at the baseline visit and the post-intervention visit, and Ecological Momentary Assessment (EMA) outcomes including pain, mood, sleep, behavior, and medication, collected up to 4 times per day during the baseline and PRT (intervention) period. Secondary outcomes include a range of state-based outcomes collected at the baseline visit and the post-intervention visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 (inclusive)
* Qualifying for Chronic Widespread Pain (CWP), as described in ICD-11 (an existing diagnosis of fibromyalgia qualifies for CWP)
* Baseline pain with an average intensity of at least 4/10 that has lasted for 3 months or longer
* If on medication that could potentially interfere with study participation or outcomes as evaluated by the study physician, stable doses of medication for 6 weeks prior to entering the study and during participation
* Living in Norway
* Fluent in Norwegian
* Normal or corrected-to-normal vision
* Access to smartphone or equivalent for use of app during study

Exclusion Criteria:

* Current comorbid acute pain condition (pain from acute illness, injury, infection, or similar in the past 3 weeks)
* Beck Depression Index (BDI) score more than 30
* Clinical high risk for suicidality (BDI short form item 7 on suicidality rated ≥ 2, or modaterate/high scores for suicidality in M.I.N.I. interview)
* Current psychological therapy for pain or mental health purposes
* Any current or past diagnosis and/or significant symptoms of psychosis-related disorders (schizophrenia, schizoaffective disorder), bipolar disorder, autism spectrum disorder, personality disorder
* Current diagnosis and/or significant symptoms of post-traumatic stress disorder (PTSD), eating disorder, substance use disorder, obsessive-compulsive disorder (OCD)
* Currently participating in other therapeutic trials
* Currently in a legal process regarding disability benefits.
* Currently pregnant
* Started an antidepressant or changed dose in the past 6 weeks
* Inability to reliably complete tasks related to the study
* Any impairment, activity or situation that in the judgement of the Study Coordinator or Principal Investigator would prevent satisfactory completion of the study protocol. This includes unreliable, or inconsistent pain scores as deemed by the principal investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Ecological Momentary Assessment (EMA) questionnaire | During baseline (6-14 days, pseudorandomized) and throughout the intervention period (4-6 weeks)
  Participants will answer EMA questions 4 times per day (morning, noon/early afternoon, afternoon, and evening) during the baseline period (6-14 days, pseudorandomized) and throughout the intervention period (4-8 weeks). Every questionnaire includes questions about current activity, affect, mood, pain, and social connectedness. The morning questionnaire includes an additional question about sleep quality, and the evening questionnaire includes additional questions about rest, feeling present, medicine use, pain-related worrying, overall pain intensity, perceived ability to manage pain, adjustment of daily activities due to pain, and avoidance of pain throughout the day. Additionaly, each individual answer a personal targeted question (evening only) formulated in collaboration with the patient with at baseline. While most questions are rated using Visual Analog Scale (VAS), some use open text (current activity, medicine), yes/no (current pain), multiple choice (pain location, rest).
Change from baseline in the Brief Pain Inventory (BPI) - Pain severity | From enrolment to the end of treatment at 4-6 weeks
  The Brief Pain Inventory is a 17-items questionnaire that assesses pain severity (0-10 Numeric Rating Scale, NRS), pain interference with activities (0-10 NRS), medication used for pain, and a body map in which the participant may mark body areas where pain is present.
Change from baseline in the Brief Pain Inventory (BPI) - Pain interference | From enrolment to the end of treatment at 4-6 weeks
  The Brief Pain Inventory is a 17-items questionnaire that assesses pain severity (0-10 Numeric Rating Scale, NRS), pain interference with activities (0-10 NRS), medication used for pain, and a body map in which the participant may mark body areas where pain is present.

SECONDARY OUTCOMES:
Change from baseline in the Pain Catastrophizing Scale (PCS) | From enrolment to the end of treatment at 4-6 weeks
  The Pain Catastrophizing Scale (PCS) is a 13 item scale that measures catastrophic thinking related to pain. The questionnaire is rated using a 0-4 Likert scale and is scored using the three subscales rumination, magnification, and helplessness, or a total sum score for all items.
Change from baseline in the Pain Coping Questionnaire - short form | From enrolment to the end of treatment at 4-6 weeks
  The Pain Coping Questionnaire (short form) is a 16-item questionnaire that is rated using a 1-5 Likert scale.
Change from baseline in the State-Trait Anxiety Inventory (State questionnaire only) | From enrolment to the end of treatment at 4-6 weeks
  The State-Trait Anxiety Inventory (STAI) consists of two similar 20-item questionnaires that measures trait-based anxiety and state-based (situational) anxiety, rated on a 1-4 Likert scale. Only the part measuring state (situational) anxiety will be used.
Change from baseline in the Generalized Anxiety Disorder Assessment (GAD-7) | From enrolment to the end of treatment at 4-6 weeks
  The GAD-7 is a 7-item scale that measures generalized anxiety, and is routinely used as a screening tool for generalized anxiety disorder. The questionnaire uses a 0-3 Likert scale.
Change from baseline in the Becks Depression Inventory II (BDI-2) | From enrolment to the end of treatment at 4-6 weeks
  The BDI-2 is a 21-item questionnaire measuring depression, using a 0-3 Likert scale
Change from baseline in the Snaith-Hamilton Pleasure Scale (SHAPS) | From enrolment to the end of treatment at 4-6 weeks
  The SHAPS measures the capacity to experience pleasure (hedonic tone) and uses a 1-4 Likert scale. A higher score indicates higher level of anhedonia.
Change from baseline in the Life Satisfaction Questionnaire (LISAT-11) | From enrolment to the end of treatment at 4-6 weeks
  The LISAT-11 is an 11-item scale measuring satisfaction with different aspects of life and uses a 1-6 Numeric Rating Scale.
Change from baseline in the PROMIS-29 | From enrolment to the end of treatment at 4-6 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS-29) is a 29-item questionnaire designed for chronic pain patients, that measures physical function, anxiety, depression, fatigue, sleep problems, ability to participate in social activities, pain interference in activities, and pain intensity.
Change from baseline in the Multidimensional Assessment of Interoceptive Awareness 2 brief version (brief MAIA-2) | From enrolment to the end of treatment at 4-6 weeks
  The brief MAIA-2 is a 24-item scale measures different aspects of interoceptive awareness using a 0-5 Numeric Rating Scale.
Change from baseline in the Perceived Stress Scale brief version | From enrolment to the end of treatment at 4-6 weeks
  The Perceived Stress Scale (brief version) is a 10-item scale measuring thoughts and feelings about stress using a 0-4 Likert Scale.
Change from baseline in the Stress Mindset Measure (SMM) | From enrolment to the end of treatment at 4-6 weeks
  The SMM is a 8-item scale measuring the extent to which an individual adopts a mindset that the effects of stress are enhancing or debilitating. It uses a 0-4 Likert Scale.
Change from baseline in the brief Existential Isolation Scale | From enrolment to the end of treatment at 4-6 weeks
  The EIS is a 6-item scale that measures social isolation as an existential experience, and uses a 0-9 Numeric Rating Scale.
Change in the Working Alliance Inventory (WAI) throughout the course of Pain Reprocessing Therapy | Up to 6 hours after every 2 PRT sessions (assessed until the last PRT session, up to 4-6 weeks after enrolment)
  The WAI is a 12-item questionnaire measuring the therapeutic alliance between a psychotherapist and a client, and is answered by the client. The WAI uses a 1-7 Likert Scale.
Life Orientation Test (LOT-R) | Baseline
  The revised Life Orientation Test (LOT-R) is a 10-item questionnaire measuring dispositional optimism and pessimism, and uses a 0-4 Likert scale, in which higher scores indicate higher dispositional optimism and lower dispositional pessimism.

OTHER OUTCOMES:
Change from baseline in the Brief Pain Inventory (BPI) - Medication | From enrolment to the end of treatment at 4-6 weeks
  The Brief Pain Inventory is a 17-items questionnaire that assesses pain severity (0-10 Numeric Rating Scale, NRS), pain interference with activities (0-10 NRS), medication used for pain, and a body map in which the participant may mark body areas where pain is present.
Change from baseline in the Brief Pain Inventory (BPI) - Body map | From enrolment to the end of treatment at 4-6 weeks
  The Brief Pain Inventory is a 17-items questionnaire that assesses pain severity (0-10 Numeric Rating Scale, NRS), pain interference with activities (0-10 NRS), medication used for pain, and a body map in which the participant may mark body areas where pain is present.

CONTACTS AND LOCATIONS:
Overall Officials: Dan-Mikael Ellingsen, PhD, Principal Investigator — Oslo University Hospital: Oslo Universitetssykehus
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data from participants who agree to have their anonymized data shared for research purposes will be made available.
Supporting Information: Study Protocol
Time Frame: From publication of the primary results until 5 years after study completion.
Access Criteria: Anonymized data and analysis code will be shared through publicly available databases such as Open Science Framework.